CLINICAL TRIAL: NCT01156051
Title: Effect of Guanfacine Extended-Release on Attention Deficit Hyperactivity Disorder (ADHD)-Associated Insomnia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: extended beyond completion date; chose to close out rather than renew IRB review
Sponsor: Children's Specialized Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Thomas Rugino, Principal Investigator, Children's Specialized Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSHTR-TR-0901; NCT01153178 (obsolete NCT alias)
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; Attention Deficit Disorder; Insomnia; Sleep Disorders
Keywords: ADHD; ADD; sleep disturbance
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Parasomnias | interventions — Guanfacine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guanfacine Extended-Release Tablets (Experimental): Guanfacine Extended-Release Tablets 1mg, 2mg, 3mg, and 4mg
  Interventions: Drug: Guanfacine extended-release tablets
- Placebo comparator (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Guanfacine extended-release tablets — Guanfacine extended-release tablets will be started at 1mg and then increased at weekly intervals to 2mg, 3mg, or 4mg as needed and as tolerated
  Other Names: Intuniv (TM), guanfacine HCl, SPD503
  Arms: Guanfacine Extended-Release Tablets
Drug: Placebo comparator — Placebo tablets identical to the experimental arm guanfacine extended-release tablets 1mg, 2mg, 3mg, 4mg, but without the active ingredient (guanfacine).
  Other Names: "sugar pill"
  Arms: Placebo comparator

SUMMARY:
This study seeks to determine, using special sleep tests (polysomnography and actigraphy) if guanfacine extended release is able to improve nighttime sleep in children with ADHD - associated insomnia while improving daytime ADHD symptoms. Male and female children with diagnosed or suspected ADHD with sleep problems (difficulty falling asleep, difficulty staying asleep, or less than expected hours of sleep) will be recruited. After obtaining informed consent and assent (when appropriate) and after discontinuation of excluded medications, children will have evaluations of his or her sleep and evaluations confirming the ADHD diagnosis. Children who successfully pass screening will be enrolled into the double-blind, placebo-controlled, randomized investigation with 50% of participants receiving guanfacine extended release and 50% of participants receiving matching placebo. Using a flexible-dose optimization design based on ADHD symptom improvement and medication tolerability, the dose will be adjusted between 1 to 4 mg over the course of four weeks. At the end of medication adjustment (week 4 or 5), ADHD questionnaires, sleep questionnaires, and sleep tests will be repeated and analyzed. The medication will be weaned over the course of the following 3-10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or female, aged 6 - 12 years with ADHD.
2. Subject must (a) be taking methylphenidate, amphetamine, or atomoxetine for treatment of ADHD with parent or subject concerns of inadequate efficacy or intolerable side effects, or (b) free of any other medication used to treat ADHD for at least 30 days at the time of the initial sleep study.
3. Subject must have repeated difficulty with sleep initiation or persistence despite attempts at adequate sleep hygiene.
4. Subject must be able to swallow tablets.

Exclusion Criteria:

1. Subject or parent/LAR is unable or unwilling to discontinue present medications used to treat ADHD.
2. Subject has a body mass index < 5th percentile for age, using the Centers for Disease Control standards reported in 2000.
3. Subject has a body weight > 176 pounds.
4. Subject has a diagnosis of Autism or Autism Spectrum Disorder.
5. Subject has other serious psychiatric diagnoses.
6. Subject has a medical condition that may require treatment with an unapproved medication, that may cause a safety concern, or that may confound outcome results
7. Subject has an excessive caffeine intake (greater than 2.5 mg/kg/d).
8. Subject has a prior problem with clonidine or guanfacine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Rugino, MD, Principal Investigator — Children's Specialized Hospital
Locations (2):
- United States (2):
  - Children's Specialized Hospital, Hamilton, New Jersey
  - Children's Specialized Hospital, Toms River, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2010 to 2012, children were referred primarily from the outpatient practice affiliated with a community based hospital dedicated to the evaluation and management of children with special needs. Four patients were referred from community pediatricians who commonly refer to the practice.
Pre-assignment Details: Medications for ADHD, that would affect sleep/alertness, or that had psychoactive properties were discontinued prior to polysomnography. Of the 35 who entered screening, 29 were enrolled. Children were disquialified for not meeting diagnostic criteria or for having disqualifying conditions (e.g., depression, heart pathology).
Groups:
- Treatment Group: Children who received (double blinded, randomized) guanfacine extended release tablets in a flexible dosing protocol, with doses ranging from 1mg to 4mg administered once daily in the morning.
- Control: Children who received a matching placebo tablet administered once daily in the morning in a flexible dosing protocol, with tablets identical to guanfacine extended release from 1mg to 4mg.
Period: Overall Study
Arm/Group | Treatment Group | Control
Started | 12 | 17
Completed | 11 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — patient not compliant with protocol | 0 | 1

BASELINE CHARACTERISTICS:
Population: 29 enrollees, but two were excluded due to (1) lost to follow up, and (2) noncompliance with the protocol.
Groups:
- Guanfacine Extended-Release Tablets: Guanfacine Extended-Release Tablets 1mg, 2mg, 3mg, and 4mg
  Guanfacine extended-release tablets: Guanfacine extended-release tablets were started at 1mg and then increased at weekly intervals to 2mg, 3mg, or 4mg as needed and as tolerated
- Placebo Comparator: Placebo control
  Placebo comparator: Placebo tablets identical to the experimental arm guanfacine extended-release tablets 1mg were started and then increased at weekly intervals to 2mg, 3mg, or 4mg as needed and as tolerated
- Total: Total of all reporting groups
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator | Total
Number analyzed (Participants) | 11 | 16 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.8) | 8.8 (1.9) | 8.9 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10 | 12 | 22
  African-American | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Polysomnographic Total Sleep Time (TST)
Description: Change in objective measures of sleep, using polysomnography
Time Frame: Baseline to last observation carried forward (after at least one week of dose stability)
Population: 29 children were enrolled, one (treatment) was lost to follow up an one (placebo) was discontinued due to noncompliance with protocol.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator
Number analyzed (Participants) | 11 | 16
minutes | -57.32 (89.17) | 31.32 (59.54)
Statistical Analysis 1: Comparison: Guanfacine Extended-Release Tablets vs Placebo Comparator; Null hypothesis: no difference in total sleep time (TST) from baseline to termination. ANOVA single measure, two-tailed, Type II analysis was completed using SPSS; Test type: Superiority or Other; p = 0.005, ANOVA

2. Secondary Outcome: Change in Baseline to Treatment ADHD-Rating Scale IV Total Score
Description: Change in baseline to treatment ADHD-Rating Scale IV (Investigator-interview ) total. This scale quantitates ADHD symptoms based on DSM-IV criteria with a minimum score of 0 and a maximum score of 54 (higher scores suggesting more ADHD symptoms). The total score is a sum of the 9 items on the ADHD Rating Scale IV inattention score and the 9 items on the ADHD Rating Scale IV hyperactivity-impulsivity score (scores for each 0-27).
Time Frame: Baseline to last observation carried forward (after at least one week of dose stability)
Population: 29 children enrolled, but two were discontinued before termination data was available: one (treatment) was lost to follow up and one (placebo) was noncompliant with the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator
Number analyzed (Participants) | 11 | 16
units on a scale | -18.27 (11.31) | -1.69 (9.16)
Statistical Analysis 1: Comparison: Guanfacine Extended-Release Tablets vs Placebo Comparator; Null hypothesis: no difference in ADHD Rating Scales - IV total scores from baseline to termination. ANOVA single measure, two-tailed, Type II analysis was completed using SPSS; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Change in Baseline to Treatment Latency to Persistent Sleep (LPS)
Description: Change in an objective measure of sleep onset, using polysomnography.
Time Frame: Baseline to last observation carried forward (after at least one week of dose stability)
Population: 29 children were enrolled; two were disqualified: one (treatment) was lost to follow-up,and one (placebo) was noncompliant with the protocol.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator
Number analyzed (Participants) | 11 | 16
minutes | 10.54 (88.44) | -19.94 (54.12)
Statistical Analysis 1: Comparison: Guanfacine Extended-Release Tablets vs Placebo Comparator; Null hypothesis: no difference in latency to persistent sleep (LPS) from baseline to termination. ANOVA single measure, two-tailed, Type II analysis was completed using SPSS; Test type: Superiority or Other; p = 0.392, ANOVA

4. Secondary Outcome: Change in Baseline to Treatment Minutes of Wake Time After Sleep Onset (WASO)
Description: Polysomnographic parameter of sleep assessing how many minutes of wakefulness occurred after sleep onset and before full morning awakening.
Time Frame: Baseline to last observation carried forward (after at least one week of dose stability)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator
Number analyzed (Participants) | 11 | 16
minutes | 21.80 (18.51) | -3.90 (17.20)
Statistical Analysis 1: Comparison: Guanfacine Extended-Release Tablets vs Placebo Comparator; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.059, ANOVA

ADVERSE EVENTS:
Arm/Group | Guanfacine Extended-Release Tablets | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 9/12 | 11/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine Extended-Release Tablets (N=12) | Placebo Comparator (N=17)
somnolence / sedation (Nervous system disorders) | 8 (8) | 1 (1) — sedation, somnolence, tired, sense of wanting to sleep
headache (Nervous system disorders) | 4 (4) | 2 (2) — headache, head pain
stomachache / abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) — stomachache, abdominal pain, abdominal discomfort
acute gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2) — infectious gastroenteritis
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — decreased appetite, anorexia, appetite decrease
inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) — inguinal hernia detected
febrile illness (Infections and infestations) | 1 (1) | 0 (0) — febrile illness, fever, acute nonspecific illness with fever
upper respiratory infection (Infections and infestations) | 3 (3) | 3 (3) — upper respiratory infection, cold, URI, coryza, stuffiness
exacerbation of allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) — allergic rhinitis, allergies, hay fever
exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — exacerbation of asthma, asthma, wheezing, cough
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — cough without asthma, cough
enuresis (Renal and urinary disorders) | 1 (1) | 0 (0) — enuresis, bedwetting, nighttime incontinence, bedwetting accidents
dizziness (Nervous system disorders) | 1 (1) | 0 (0) — dizziness, lightheadedness
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — chest pain not of cardiac origin, chest wall tenderness, costochondritis
oral pain due to loose teeth (General disorders) | 1 (1) | 0 (0) — oral pain due to loose teeth (developmental in nature)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — dermatitis, rash, contact dermatitis
stuttering (Psychiatric disorders) | 0 (0) | 1 (1) — stuttering

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No